CLINICAL TRIAL: NCT03467074
Title: Association of Genetic Polymorphisms in the Interferon-λ Signaling Cascade and Immune Response After Vaccination
Brief Title: Role of Interferon-λ and Vaccine Response
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-141; me15Egli
Record Dates: First submitted 2018-03-06; First posted 2018-03-15 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Vaccine Response Impaired; Allogeneic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: influenza A/B vaccine — Regardless of the study enrollment, a two-time influenza vaccination at the start of the flu season is recommended every 4 weeks for all patients after stem cell transplantation. The vaccine is a trivalent inactivated non-adjuvanted influenza virus vaccine containing two influenza A viruses: pandemic H1N1, and H3N2, and an influenza B virus

SUMMARY:
The following observational study will investigate whether the vaccine response (antibodies, T and B cells) after allogeneic stem cell transplantation is influenced by genetic polymorphisms in the interferon lambda signal.

DETAILED DESCRIPTION:
The research project deals with one of the most important virological preventive measures after stem cell transplantation: vaccination against influenza viruses. Patients with allogeneic stem cell transplantation may experience serious complications of influenza and are at higher risk for inadequate response to the vaccine. The research project will make it possible, in a translational-medical orientation, to investigate the exact influence of genetic polymorphisms of the Interferon (IFN)-λ signalling cascade on the immune response after vaccination. This knowledge will make it possible to identify high-risk patients for a poor vaccination response before vaccination and to personalize the current vaccination strategy (intra-muscular injection), e.g. by subcutaneous vaccination, repeated administration of the vaccine or vaccine with adjuvants.

ELIGIBILITY:
Inclusion Criteria:

* held allogeneic stem cell transplantation over 1 year ago

Exclusion Criteria:

* Known vaccine intolerance (e.g. Protein allergy or severe vaccine-associated side effects, e.g. Guillian Barré syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after allogeneic stem cell transplantation, which are in control at the University Hospital Basel, Cantonal Hospital Aarau, Lucerne Cantonal Hospital, University Hospital Zurich, Inselspital Bern or the Regional Hospital Bellinzona.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Peripheral Blood Mononuclear Cells (PBMCs) in blood before vaccination | Change from baseline PBMCs at day 60
  Before vaccination, antibody titers for each influenza virus contained in the vaccine (Influenza A pH1N1, Influenza A H3N2 and Influenza B) are determined from the serum by means of a hemagglutination inhibition assay (HIA titer)
Peripheral Blood Mononuclear Cells (PBMCs) in blood after vaccination | Change from baseline PBMCs at day 60
  after vaccination, antibody titers for each influenza virus contained in the vaccine (Influenza A pH1N1, Influenza A H3N2 and Influenza B) are determined from the serum by means of a hemagglutination inhibition assay (HIA titer)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD MD, Principal Investigator — Department of Clinical Microbiology
Locations (1):
- Department of Clinical Microbiology, Basel, Switzerland

REFERENCES:
- [Derived] Linnik J, Syedbasha M, Kaltenbach HM, Vogt D, Hollenstein Y, Kaufmann L, Cantoni N, Ruosch-Girsberger S, Muller AMS, Schanz U, Pabst T, Stussi G, Weisser M, Halter J, Stelling J, Egli A. Association of Host Factors With Antibody Response to Seasonal Influenza Vaccination in Allogeneic Hematopoietic Stem Cell Transplant Patients. J Infect Dis. 2022 Apr 19;225(8):1482-1493. doi: 10.1093/infdis/jiab391. PMID 34415049